CLINICAL TRIAL: NCT02990988
Title: Microbiome of Donor Iron Deficient Study (DIDS)
Brief Title: Microbiome of Donor Iron Deficient Study
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAR1265
Record Dates: First submitted 2016-12-09; First posted 2016-12-13 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Iron Deficiency
Keywords: Blood donation; Iron repletion; Transfusion
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stool collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Iron repletion: Subjects participating in the associated study under the Iron Repletion arm will also provide stool collection and answers to questionnaire and diet diary.
- Placebo: Subjects participating in the associated study under the Placebo arm will also provide stool collection and answers to questionnaire and diet diary.

SUMMARY:
The goal of this pilot study is to test whether the microbiome is affected by intravenous iron repletion.

DETAILED DESCRIPTION:
The colonic microbiome, the community of bacteria living in our gut, is essential in human health and disease. Iron is an essential nutrient for both bacteria and humans. In the United States, of the donors who provided the ~15 million units of red blood cells that were collected for transfusion, 69% were repeat donors. Although iron deficiency is surprisingly prevalent in first-time donors, its prevalence is even higher in these particularly altruistic frequent donors, (i.e., up to 49% and 66% of male and female repeat donors, respectively), manifested as iron depletion or iron-deficient erythropoiesis. Iron deficiency from blood donation is associated with fatigue, restless leg syndrome, decreased physical endurance and work capacity, and impaired concentration, attention, and other neurocognitive functions; however, these conclusions are not based on definitive studies and have not yet changed blood donation policy. The goal is to conduct a prospective, double-blind, randomized controlled trial, recruiting 60 healthy regular donors who meet donation standards, while exhibiting iron-deficient erythropoiesis by laboratory test criteria. In this ancillary study, we will determine what effect donor iron deficiency and IV iron repletion have on the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Current participant of the associated randomized controlled trial conducted at Columbia University Medical Center (therefore invited to participate in this optional ancillary study).

Exclusion Criteria:

* Not a current participant of the associated randomized controlled trial conducted at Columbia University Medical Center.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with iron deficiency from blood donation will be recruited over 5 years in the associated randomized controlled trial conducted at Columbia University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2017-01; Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Change in overall diversity of fecal flora | Baseline, 5-days, 4-weeks, 5 months
  Stool samples will be collected and processed.
Change in fecal indoles | Baseline, 5-days, 4-weeks, 5 months
  Indole concentrations measured in fecal samples
Change in fecal iron | Baseline, 5-days, 4-weeks, 5 months
  Iron concentrations measured in fecal samples

SECONDARY OUTCOMES:
Mean Bray-Curtis indices | Baseline, 5-days, 4-weeks, 5 months
  Calculation of Bray-Curtis index will determine the relative abundance of specific taxa (e.g., Firmicutes, Bacteroidetes, Proteobacteria) for each subject. Means (of the differences in %) and standard deviations will be calculated for all comparisons, and a multivariable generalized estimating equations (GEE) model will be used to test for significance.

CONTACTS AND LOCATIONS:
Overall Officials: Eldad Hod, MD, Principal Investigator — Associate Professor of Pathology and Cell Biology, Dept of Pathology&Cell Biology
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith GA, Fisher SA, Doree C, Roberts DJ. A systematic review of factors associated with the deferral of donors failing to meet low haemoglobin thresholds. Transfus Med. 2013 Oct;23(5):309-20. doi: 10.1111/tme.12046. Epub 2013 Jul 5. PMID 23829880
- [Background] Newman B. Iron depletion by whole-blood donation harms menstruating females: the current whole-blood-collection paradigm needs to be changed. Transfusion. 2006 Oct;46(10):1667-81. doi: 10.1111/j.1537-2995.2006.00969.x. No abstract available. PMID 17002622
- [Background] Bialkowski W, Bryant BJ, Schlumpf KS, Wright DJ, Birch R, Kiss JE, D'Andrea P, Cable RG, Spencer BR, Vij V, Mast AE. The strategies to reduce iron deficiency in blood donors randomized trial: design, enrolment and early retention. Vox Sang. 2015 Feb;108(2):178-85. doi: 10.1111/vox.12210. Epub 2014 Dec 3. PMID 25469720
- [Background] Cable RG, Glynn SA, Kiss JE, Mast AE, Steele WR, Murphy EL, Wright DJ, Sacher RA, Gottschall JL, Tobler LH, Simon TL; NHLBI Retrovirus Epidemiology Donor Study-II (REDS-II). Iron deficiency in blood donors: the REDS-II Donor Iron Status Evaluation (RISE) study. Transfusion. 2012 Apr;52(4):702-11. doi: 10.1111/j.1537-2995.2011.03401.x. Epub 2011 Oct 24. PMID 22023513
- [Background] Brittenham GM. Iron deficiency in whole blood donors. Transfusion. 2011 Mar;51(3):458-61. doi: 10.1111/j.1537-2995.2011.03062.x. No abstract available. PMID 21388389